CLINICAL TRIAL: NCT01347736
Title: Scrambler Therapy for the Treatment of Chronic Zoster Pain
Brief Title: Scrambler Therapy in Treating Chronic Pain in Patients With Rash From Varicella Zoster Virus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC10CE; NCI-2011-00338 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC10CE (Other: Mayo Clinic Cancer Center); 11-00531 (Other: Mayo Clinic IRB); NCI-2011-00338 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-03-30; First posted 2011-05-04 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-02

CONDITIONS: Dermatologic Complications; Pain; Viral Infection
MeSH Terms: conditions — Pain; Virus Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pain therapy) (Experimental): Patients undergo scrambler therapy for approximately 30 minutes. Treatment continues for 10 days in the absence of pain progression or unacceptable toxicity.
  Interventions: Other: scrambler therapy; Other: questionnaire administration; Procedure: dermatologic complications management/prevention

INTERVENTIONS:
Other: scrambler therapy — Undergo scrambler therapy
Other: questionnaire administration — Ancillary studies
Procedure: dermatologic complications management/prevention — Undergo scrambler therapy
  Other Names: complications management/prevention, dermatologic; management/prevention, dermatologic complications

SUMMARY:
This pilot clinical trial studies how well scrambler therapy works treating chronic pain in patients with rash from varicella zoster virus infection. Scrambler therapy may help relieve pain from a rash caused by varicella zoster virus infection

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore whether we can decrease post-herpetic neuralgia (PHN) pain with scrambler therapy.

OUTLINE: Patients undergo scrambler therapy for approximately 30 minutes. Treatment continues for 10 days in the absence of pain progression or unacceptable toxicity. After the completion of study treatment, patients are followed up for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pain of >= 1 month (30 days) duration attributed to zoster, for which the patient wants intervention
* Pain at least a four out of ten problem during the prior week, on a 0-10 scale where zero was no problem and ten was the worst possible problem
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) = 0, 1, or 2
* Life expectancy >= 3 months (90 days)
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide informed written consent

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown
* Pregnant women
* Patients with implantable drug delivery systems, e.g. Medtronic Synchromed
* Patients with heart stents or metal implants such as pacemakers, automatic defibrillators, aneurysm clips, vena cava clips and skull plates; (metal implants for orthopedic repair, e.g. pins, clips, plates, cages, joint replacements are allowed as are central venous access devices)
* Patients with a history of myocardial infarction or ischemic heart disease within the past six months
* Patients with history of epilepsy, brain damage, use of anti-convulsants for seizure prevention, symptomatic brain metastases; Note: anti-convulsant use is allowed for neuropathy and heart failure (HF) if on a stable dose
* Other identified causes of pain in the area that was affected by herpes zoster
* Skin conditions such as open sores that would prevent proper application of the electrodes
* Other medical or other condition(s) that in the opinion of the investigators might compromise the objectives of the study
* Prior treatment with Calmare MC-5A therapy
* Patient initiation of a new analgesic treatment within 7 days prior to initiation of protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-11-07 (Actual); Study Completion 2014-11-07 (Actual)

PRIMARY OUTCOMES:
Change in pain on a 0-10 numerical rating scale. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States